CLINICAL TRIAL: NCT04583436
Title: Efficacy and Safety Comparison of the Open (Femoral-popliteal Distal Bypass by Synthetic Vascular Graft) and Endovascular (Recanalization With Angioplasty and Stenting With Biomimetic Interwoven Nitinol Stent) Surgical Methods for the Treatment of Long Atherosclerotic Lesions of the Femoral-popliteal Segment Below the Knee, TASC D in Patients With Critical Limb Ischemia
Brief Title: Efficacy and Safety Comparison of the Open and Endovascular Surgical Methods for the Treatment of Long Atherosclerotic Lesions of the Femoral-popliteal Segment Below the Knee, TASC D in Patients With Critical Limb Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sosudi1
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Atherosclerotic Ischemic Disease; Critical Limb Ischemia; Superficial Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: intervowen biomimetic nitinol stent; TASC D; femoro-popliteal distal bypass; Critical limb ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Conversion to Open Surgery

STUDY DESIGN:
Intervention Model Description: Group 1: Femoropopliteal distal bypass with a synthetic ePTFE graft; Group 2: Recanalization of occlusion of the arteries of the femoropopliteal segment below the knee joint with angioplasty and stenting with a biomimetic intervowen nitinol stent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular recanalization (Experimental): Recanalization with angioplasty and stenting: Under local anesthesia, a standard endovascular approach is performed and the affected arterial segment is visualized. Perform transluminal or subintimal recanalization of the occluded segment of the arteries with a hydrophilic guide wire. Next, balloon angoplasty of the recanalized segment is performed. After control angiography, a biomimetic braided nitinol stent is placed throughout the lesion.
  n=45
  Interventions: Device: Endovascular recanalization
- Open surgery (Active Comparator): Femoropopliteal distal bypass with a synthetic ePTFE graft: Under general anesthesia, 2 standard open surgical approaches are performed: one to the common femoral artery, superficial femoral artery and deep femoral artery; the second - to the third portion of the popliteal artery, the tibioperoneal trunk and the anterior tibial artery. After systemic heparinization, clamps are applied to the arteries. A longitudinal arteriotomy of the popliteal artery is performed, and a distal end-to-side anastomosis is formed between the artery and the graft. Next, the graft is passed into the groin wound. Longitudinal arteriotomy of the common femoral artery. A proximal end-to-side anastomosis is formed between the shunt and the common femoral artery. Clamps are removed from arteries, blood flow is started, surgical hemostasis, wound drainage, layer-by-layer wound closure is performed.
  n=45
  Interventions: Other: Open surgery

INTERVENTIONS:
Device: Endovascular recanalization — Recanalization with angioplasty and stenting: Under local anesthesia, a standard endovascular approach is performed and the affected arterial segment is visualized. Perform transluminal or subintimal recanalization of the occluded segment of the arteries with a hydrophilic guide wire. Next, balloon angoplasty of the recanalized segment is performed. After control angiography, a biomimetic braided nitinol stent is placed throughout the lesion.
  Arms: Endovascular recanalization
Other: Open surgery — Femoropopliteal distal bypass with a synthetic ePTFE graft: Under general anesthesia, 2 standard open surgical approaches are performed: one to the common femoral artery, superficial femoral artery and deep femoral artery; the second - to the third portion of the popliteal artery, the tibioperoneal trunk and the anterior tibial artery. After systemic heparinization, clamps are applied to the arteries. A longitudinal arteriotomy of the popliteal artery is performed, and a distal end-to-side anastomosis is formed between the artery and the graft. Next, the graft is passed into the groin wound. Longitudinal arteriotomy of the common femoral artery. A proximal end-to-side anastomosis is formed between the shunt and the common femoral artery. Clamps are removed from arteries, blood flow is started, surgical hemostasis, wound drainage, layer-by-layer wound closure is performed.
  Arms: Open surgery

SUMMARY:
This is prospective, randomized study. The main objective of the study is to compare the clinical efficacy and safety of two therapies for the treatment of prolonged atherosclerotic lesions of the arteries of the femoropopliteal segment below the knee, TASC II type D - femoropopliteal distal bypass with a synthetic ePTDE-grafts and recanalization with angioplasty and stenting using a biomimetic intervowen nitinol stent in patients with symptomatic peripheral arterial disease after 24 months. Secondary objectives are to identify predictors of restenosis and occlusions of the operated segment and compare the quality of life of patients after the procedure.

DETAILED DESCRIPTION:
Steno-occlusive lesion of the superficial femoral and popliteal artery is observed from 2.5% to 14.5% (National guidelines for the management of patients with vascular arterial pathology, Russian Consensus Document, 2010) of patients in different age groups. The standard technique of autovenous femoral-femoral or femoral-popliteal bypass surgery has shown its five-year effectiveness in 66-73.7% of patients (Remote endarterectomy versus supragenicular bypass surgery for long occlusions of the superficial femoral artery: Medium-term results of a randomized controlled trial (The REVAS trial ). by Suzanne S. Gisbertz, Rudolf P. Tutein Nolthenius, Gert Jan De Borst, Lyckle Van Der Laan, Tim Th C Overtoom, Frans L. Moll, Jean Paul PM De Vries 2010). However, these results are significantly impaired by femoral-popliteal bypass grafting below the knee joint, or femoral-tibial revascularization. In this position, five-year patency is 33-50% (Johnson WC, Lee KK A comparative evaluation of polytetra-fluoroethylene, umbilical vein, and saphenous vein bypass grafts for femoral-popliteal above-knee revascularization: a prospective randomized Department of Veterans Affairs cooperative study. J. Vasc. Surg). Patients whose own vein was previously used for coronary artery bypass grafting or has a small diameter and extensive lateral branches are also very problematic for surgery. At the same time, in patients with relatively compensated chronic ischemia of the lower extremities (CLI category 2-3 according to the Rutherford classification) and the absence of autologous material for shunting, it is possible to continue with optimal drug therapy. In the case of critical lower limb ischemia (category 4-6 according to the Rutherford classification), revascularization is indicated in order to preserve the limb (National guidelines for the diagnosis and treatment of diseases of the lower limb arteries, Section 7, pp. 59-61. Moscow, 2019). A common operation of percutaneous transluminal angioplasty with stenting of these arteries allows you to restore blood flow through your own arteries. However, with physiological flexion and extension of the hip and knee joints, there is a pronounced deformation of the stented popliteal and superficial femoral arteries both in the axial and angular directions. This is accompanied by breakage of the stents, or their restenosis and thrombosis. So, according to a number of authors, the two-year incidence of stent breakages in the superficial femoral artery ranges from 20% to 46% (Duda SH, Bosiers M, Lammer J, et al. Drug-eluting and bare nitinol stents for the treatment of atherosclerotic lesions in the superficial femoral artery: Long-term results from the SIROCCO trial. J Endovasc Ther 2006; 13: 701-710), and the frequency of restenosis and occlusions from 21.8% to 53.3% (Laird JR, Katzen BT, Scheinert D, et al. Nitinol stent implantation vs. balloon angioplasty for lesions in the superficial femoral and proximal popliteal arteries of patients with claudication: Three-year follow-up from the RESILIENT randomized trial. J Endovasc Ther 2012; 19: 1-9).

One of the possible solutions to the problem of stent breakage in the femoral-popliteal position is a modified method of their manufacture by braiding from nitinol wire. Pilot two-year studies with braided stents have indeed shown resistance to breakage in this position. Moreover, the frequency of restenosis was observed in 27.2% of patients (M. Werner, A. Paetzold, U. Banning-Eichenseer, S. Scheinert, M. Piorkowski, M. Ulrich, Y. Bausback, S. Bräunlich, A. Schmidt, D. Scheinert. Treatment of complex atherosclerotic femoropopliteal artery disease with a self-expanding interwoven nitinol stent: midterm results from the Leipzig SUPERA 500 registry // EuroIntervention 2014; March 2014).

At the same time, a recent study, where the authors studied the effectiveness of stenting of long lesions (200 mm or more) of the femoral-popliteal segment with BRM stents, showed unsatisfactory indicators (45%) of the patency of the stented segment within 2 years (Lin Y, Tang X, Fu W, Kovach R, George JC, Guo D. Stent fractures after superficial femoral artery stenting: risk factors and impact on patency. Journal of Endovascular Therapy. 2015 Jun; 22 (3): 319-26). This fact proves the need for a comparative study on such a cohort of patients using a interwoven nitinol stent, devoid of some of the disadvantages of usual BRM stents (as described above), which will improve the efficiency of this procedure both in the early and late postoperative period. Recently published by authors (Garcia L, Jaff MR, Metzger C, Sedillo G, Pershad A, Zidar F, Patlola R, Wilkins RG, Espinoza A, Iskander A, Khammar GS Wire-interwoven nitinol stent outcome in the superficial femoral and proximal popliteal arteries: twelve-month results of the SUPERB trial) the results of the effectiveness of such a procedure within 12 months, but with a shorter average length of the lesion (78.1 mm) showed encouraging results (the primary 12-month patency was 78.9%), which gives hope for good results even with long lesions.

Technology description:

Recanalization with angioplasty and stenting: Under local anesthesia, a standard endovascular approach is performed and the affected arterial segment is visualized. Perform transluminal or subintimal recanalization of the occluded segment of the arteries with a hydrophilic guide wire. Next, balloon angoplasty of the recanalized segment is performed. After control angiography, a biomimetic braided nitinol stent is placed throughout the lesion.

Drug therapy includes pre-procedure aspirin (160-300 mg / day), starting at least one day before, and intra-procedure heparin (100 U / kg body weight intravenously). After the procedure, all patients are prescribed aspirin (100 mg per day) for a long time and clopidogrel (75 mg per day) for 3 months.

Femoropopliteal distal bypass with a synthetic ePTFE graft: Under general anesthesia, 2 standard open surgical approaches are performed: one to the common femoral artery, superficial femoral artery and deep femoral artery; the second - to the third portion of the popliteal artery, the tibioperoneal trunk and the anterior tibial artery. After systemic heparinization, clamps are applied to the arteries. A longitudinal arteriotomy of the popliteal artery is performed, and a distal end-to-side anastomosis is formed between the artery and the graft. Next, the graft is passed into the groin wound. Longitudinal arteriotomy of the common femoral artery. A proximal end-to-side anastomosis is formed between the shunt and the common femoral artery. Clamps are removed from arteries, blood flow is started, surgical hemostasis, wound drainage, layer-by-layer wound closure is performed.

Drug therapy includes pre-procedure aspirin (160-300 mg / day), starting at least one day before, and intra-procedure heparin (100 U / kg body weight intravenously). After the procedure, all patients are prescribed aspirin (75-100 mg per day) for a long time.

The aim of the study: to evaluate the efficacy and safety of two methods of treatment of prolonged atherosclerotic lesions of the arteries of the femoropopliteal segment below the knee within 24 months after treatment.

Research objectives:

* Evaluate the effectiveness of two methods of treatment of prolonged atherosclerotic lesions of the arteries of the femoropopliteal segment below the knee joint after 24 months (primary patency, primary-assisted patency, secondary patency, TLR, MALE);
* Evaluate the safety of two methods of treatment of prolonged atherosclerotic lesions of the arteries of the femoral-popliteal segment below the knee joint in the early postoperative period (hematoma, peripheral neuropathy, purulent-infectious complications of the surgical access area) and after 24 months (MACE)
* Assess the quality of life in patients after surgery after 1, 12 and 24 months;
* Assess prognostic factors for adverse outcomes.

Population:

Male and female patients > 18 years old with diagnosed atherosclerotic occlusive lesion of the femoropopliteal segment below the knee (TASC II type D) requiring surgical correction, recruited in accordance with the inclusion / exclusion criteria.

Sample Size:

The literature data review of studies on endovascular (using intervowen biomimetic nitinol stents) and open revascularization (femoral-popliteal distal bypass) arteries of the infrainguinal segment shown (Scheinert, D., Grummt, L., Piorkowski, M., Sax, J., Scheinert, S., Ulrich, M., ... Schmidt, A. (2011). A Novel Self-Expanding Interwoven Nitinol Stent for Complex Femoropopliteal Lesions: 24-Month Results of the SUPERA SFA Registry. Journal of Endovascular Therapy, 18 (6), 745-752. Https://doi.org/10.1583/11-3500.1), that 2-year primary patency after endovascular revascularization using a biomimetic intervowen nitinol stent was 76.1 ± 4.5%. At the same time, the two-year primary patency after femoropopliteal distal bypass surgery using an artificial ePTFE grafts is about 40% (Eickhoff JH, Broomé A, Ericsson BF, Hansen HJ, Kordt KF, Mouritzen C, Kvernebo K, Norgren L, Rostad H, Trippestad A. Four years' results of a prospective, randomized clinical trial comparing polytetrafluoroethylene and modified human umbilical vein for below-knee femoropopliteal bypass. Journal of vascular surgery. 1987 Nov 1; 6 (5): 506-11.). Given these data, a GPower analysis was performed to calculate the sample size for a study power of 80%. The sample size is 82 patients. Taking into account possible losses, it is planned to recruit 90 patients (45 in each group) with diagnosed atherosclerotic occlusive lesion of the femoropopliteal segment below the knee joint (type D according to TASC II), with chronic ischemia of the lower extremities of 3-6 categories according to Rutherford. After patients have been screened according to the inclusion / exclusion criteria, as well as voluntary written informed consent to participate in the study, randomization (envelope method) will be performed to include the patient in a particular group.

Inclusion citeria:

* Adults patients (>18 years old);
* Critical limb ischemia (4-6 Rutherford category)
* Atherosclerotic occlusive lesion of the arteries of the femoropopliteal segment below the knee joint, classified by TASC II as type D, confirmed by computed tomography or arteriography;
* De Novo lession;
* Patient consent;
* Lack of suitable autologous shunting material (GSV)

Exclusion criteria:

* Juvenile patient (< 18 years old);
* Pregnancy;
* Asymptomatic lession;
* Acute ischemia;
* Previous treatment on the target lession;
* Non-atherosclerotic lession;
* Severe comorbidity with a life expectancy - less than 2 years;
* Contraindications to antiplatelet therapy;
* Patient participation in another clinical trial;
* Patient refusal to participate in the study;
* Availability of suitable autologous bypass material.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (>18 years old);
* Critical limb ischemia (4-6 Rutherford category);
* Atherosclerotic occlusive lesion of the arteries of the femoropopliteal segment below the knee joint, classified by TASC II as type D, confirmed by computed tomography or arteriography;
* De Novo lession;
* Patient consent;
* Lack of suitable autologous shunting material (GSV)

Exclusion Criteria:

* Juvenile patient (< 18 years old);
* Pregnancy;
* Asymptomatic lession;
* Acute ischemia;
* Previous treatment on the target lession;
* Non-atherosclerotic lession;
* Severe comorbidity with a life expectancy - less than 2 years;
* Contraindications to antiplatelet therapy;
* Patient participation in another clinical trial;
* Patient refusal to participate in the study;
* Availability of suitable autologous bypass material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 24 months
  Primary patency was defined as absence of occlusion or flow-limiting stenosis (peak systolic velocity [PSV] ratio >2.5) of the treated segment including 1 cm proximal and distal of the anastomosis
Primary assisted patency | 24 months
  Primary assisted patency was defined as a secondary procedure is performed to prevent failure (i.e., in a flow-limiting stenosis [PSV ratio >2.5] in a still-patent segment of stent or bypass, including the anastomoses
Secondary patency | 24 months
  Secondary patency was defined as a secondary procedure performed for graft or stent occlusion in an afterward patent vessel.

SECONDARY OUTCOMES:
MALE | 24 months
  Major adverce limb events (untreated loss of patency, reintervention on the index arterial segment, or amputation of the index limb).
Safety of the method of surgical treatment in the early postoperative period | 30 days
  (hematoma of the surgical access area, peripheral neuropathy, purulent-infectious complications of the surgical access area)
MACE | 24 months
  MACE defined as stroke, myocardial infarction, or death
Assessment of the quality of life in patients after surgical treatment | 24 months
  SF 36 questionary

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin National Medical Research Center Ministry of healthcare of Russia, Novosibirsk, Novosibirsk Area, Russia